CLINICAL TRIAL: NCT00464646
Title: A Phase II Clinical Trial of Epirubicin Plus Cyclophosphamide Followed by Docetaxel Plus Trastuzumab and Bevacizumab Given as Neoadjuvant Therapy for HER2-Positive Locally Advanced Breast Cancer or Given as Adjuvant Therapy for HER2-Positive Pathologic Stage III Breast Cancer
Brief Title: Therapy With Bevacizumab (BEV), Epirubicin, and Cyclophosphamide Followed by Docetaxel Plus Trastuzumab and BEV Given as Neoadjuvant or Adjuvant Therapy for Women With Locally Advanced HER2 Positive Invasive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Genentech, Inc. (Industry); International Drug Development Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FB-5
Record Dates: First submitted 2007-04-19; First posted 2007-04-23 (Estimated); Results first posted 2012-09-26 (Estimated); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: NSABP; Epirubicin; Cyclophosphamide; Docetaxel; Trastuzumab; Bevacizumab; Neoadjuvant Therapy; HER2; Locally Advanced Breast Cancer; Adjuvant Therapy; Pathologic Stage III Breast Cancer; Inflammatory Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Epirubicin; Cyclophosphamide; Docetaxel; Trastuzumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): * Cohort A: Women with unresected locally advanced breast cancer (clinical Stage IIIA, IIIB, and IIIC)
  * Cohort B: Women with resected pN2 or pN3 (pathologic Stage III) breast cancer
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Trastuzumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Epirubicin — Both Cohorts: Epirubicin 90 mg/m2 IV every 21 days x 4 cycles
  Other Names: Ellence
Drug: Cyclophosphamide — Both Cohorts: Cyclophosphamide 600 mg/m2 IV every 21 days x 4 cycles
Drug: Docetaxel — Both Cohorts: Docetaxel 100 mg/m2 IV on Day 1 every 21 days x 4 cycles
  Other Names: Taxotere
Drug: Trastuzumab — Cohort A: Pre-op therapy - 4 mg/kg IV first dose, then subsequent doses at 2 mg/kg IV weekly (16+ weeks) until 1-7 days prior to surgery. Post-operative therapy (beginning no sooner than 28 days after surgery and continuing every 3 weeks x 13 doses) - 8 mg/kg IV first post-op dose, then subsequent doses at 6 mg/kg IV
  Cohort B: 4 mg/kg IV first dose, then subsequent doses at 2 mg/kg IV weekly on days 1, 8, and 15. Three (3) weeks after last dose of docetaxel, 6 mg/kg IV and continuing every 3 weeks x 13 doses
  Other Names: Herceptin
Drug: Bevacizumab — Cohort A: Cycles 1-4, 15 mg/kg IV on day 1 of cycle 4 only; Cycles 5-7, 15 mg/kg IV on day 1 every 21 days x 3 cycles; post-operative therapy (beginning no sooner than 28 days after surgery), 15 mg/kg IV every 3 weeks x 13 doses
  Cohort B: Cycles 5-8, 15 mg/kg IV on day 1 every 21 days x 4 cycles; beginning 3 weeks after last dose of docetaxel, 15 mg/kg IV every 3 weeks x 13 doses
  Other Names: Avastin

SUMMARY:
The main purpose is to learn if adding bevacizumab to standard chemotherapy and trastuzumab to treat HER2-positive breast cancer will affect heart function. This study will evaluate:

* How bevacizumab, given with chemotherapy, and then bevacizumab given with trastuzumab after surgery, will affect breast tumors
* Side effects from adding bevacizumab to chemotherapy and trastuzumab
* Whether adding bevacizumab to chemotherapy and trastuzumab for breast cancer will affect the heart
* If receiving bevacizumab will have any effect on how patients recover from surgery

DETAILED DESCRIPTION:
NSABP FB-5 is a Phase II study for women with HER2-positive invasive breast cancer evaluating a regimen of epirubicin plus cyclophosphamide followed by docetaxel plus trastuzumab and bevacizumab in two patient cohorts:

* Cohort A: Women with unresected locally advanced breast cancer (clinical Stage IIIA, IIIB, and IIIC)
* Cohort B: Women with resected pN2 or pN3 (pathologic Stage III) breast cancer.

The primary aims of the study are to determine the rate of cardiac events for all patients and the pCR rate in the breast and axillary lymph nodes for Cohort A. Cardiac events will be defined as NYHA Class III/IV congestive heart failure and cardiac death. For Cohort A, secondary aims of the study include determining the rate of pCR in the breast and the cCR rate following the neoadjuvant therapy. The secondary aims also include determining the value of the regimen in improving 5-year RFS and 5-year OS and determining the non-cardiac toxicities of the regimen in all patients.

Patients in Cohort A will receive neoadjuvant therapy consisting of epirubicin plus cyclophosphamide (EC) every 21 days for 4 cycles plus bevacizumab given on Day 1 of Cycle 4 only, followed by docetaxel every 21 days for 4 cycles plus bevacizumab every 21 days for the initial 3 cycles. Patients will also receive weekly trastuzumab beginning with the first cycle of docetaxel and continuing until 1-7 days before surgery. Patients will then have breast surgery (lumpectomy or mastectomy) with axillary staging. Approximately 4-6 weeks following surgery, bevacizumab and trastuzumab will resume and continue every 3 weeks for 13 doses to complete one year of targeted therapy.

Patients in Cohort B will receive adjuvant therapy consisting of EC every 21 days for 4 cycles followed by docetaxel every 21 days for 4 cycles. Beginning with the first cycle of docetaxel, patients will also receive bevacizumab every 21 days for 4 cycles and weekly trastuzumab until 3 weeks after the last docetaxel dose. Beginning 3 weeks after the last dose of docetaxel, both bevacizumab and trastuzumab will then be given every 3 weeks for 13 doses to complete 1 year of targeted therapy.

Cardiac monitoring will be conducted for both cohorts. For Cohort A, LVEF assessments will be conducted at baseline, post-EC, 2-4 weeks following surgery (about 6 months from study entry), and 9, 12, 15, and 18 months from study entry. For Cohort B, LVEF assessments will be conducted at baseline, post-EC, and 6, 9, 12, 15, and 18 months from study entry. The preferred method for LVEF assessment is 2-D echocardiogram; however, LVEF assessment by MUGA scan is permitted.

Patient follow-up will continue for 5 years following study entry.

The FB-5 sample size is 105 patients.

ELIGIBILITY:
Inclusion Criteria:

Conditions for eligibility for patients with LABC (Cohort A):

* The diagnosis of invasive adenocarcinoma of the breast must have been made by core needle biopsy or limited incisional biopsy.
* Patients must have clinical Stage IIIA, IIIB, or IIIC disease with a mass in the breast or axilla that is greater than or equal to 2.0 cm measured by clinical exam, unless the patient has inflammatory breast carcinoma, in which case measurable disease is not required.

Conditions for eligibility for patients with resected Stage III breast cancer (Cohort B)

* Patients must have undergone either a total mastectomy or a lumpectomy.
* Patients must have completed one of the following procedures for evaluation of pathologic nodal status.

  * Sentinel lymphadenectomy followed by removal of additional non-sentinel lymph nodes, or
  * Axillary lymphadenectomy without SN isolation procedure.
* The interval between the last surgery (for breast cancer treatment or staging) and study entry must be no more than 84 days.
* By pathologic evaluation, ipsilateral nodes must be pN2 or pN3.
* For patients who undergo lumpectomy, the margins of the resected specimen must be histologically free of invasive tumor and DCIS as determined by the local pathologist. If pathologic examination demonstrates tumor at the line of resection, additional operative procedures may be performed to obtain clear margins. If tumor is still present at the resected margin after re-excision(s), the patient must undergo total mastectomy to be eligible. (Patients with margins positive for LCIS are eligible without additional resection.)
* For patients who undergo mastectomy, margins must be free of gross residual tumor. Patients with microscopic positive margins are eligible.

Conditions for patient eligibility (ALL patients)

* The patient must have consented to participate and must have signed and dated an IRB-approved consent form that conforms to federal and institutional guidelines.
* Patients must be female.
* The patient must be greater than or equal to 18 years old.
* The patient's ECOG performance status must be 0 or 1.
* The tumor must be invasive adenocarcinoma of the breast on histologic examination.
* The breast cancer must be determined to be HER2-positive prior to study entry. Assays performed using FISH require gene amplification. Assays using IHC require a strongly positive (3+) staining score.
* At the time of study entry, blood counts must meet the following criteria:

  * Absolute neutrophil count (ANC) must be greater than/equal to 1200/mm3.
  * Platelet count must be greater than/equal to 100,000/mm3.
  * Hemoglobin must be greater than/equal to 10 g/dL.
* The following criteria for evidence of adequate hepatic function must be met:

  * total bilirubin must be less than/equal to ULN for the lab unless the patient has a grade 1 bilirubin elevation (greater than ULN to 1.5 x ULN) due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and
  * alkaline phosphatase must be less than 2.5 x ULN for the lab; and
  * AST must be less than/equal to 1.5 x ULN for the lab.
  * Alkaline phosphatase and AST may not both be greater than the ULN. For example, if the alkaline phosphatase is greater than the ULN but less than/equal to 2.5 x ULN, then the AST must be less than/equal to the ULN. If the AST is greater than the ULN but less than/equal to 1.5 x ULN, then the alkaline phosphatase must be less than/equal to ULN.
* Patients with AST or alkaline phosphatase greater than ULN are eligible for inclusion in the study if liver imaging (CT, MRI, or PET scan) does not demonstrate metastatic disease, and has adequate hepatic function.
* Patients with either skeletal pain or alkaline phosphatase that is greater than ULN but less than/equal to 2.5 x ULN are eligible for inclusion in the study if a bone scan or PET scan does not demonstrate metastatic disease. Patients with suspicious findings on bone scan or PET scan are eligible if suspicious findings are confirmed as benign by x-ray, MRI, or biopsy.
* Serum creatinine less than/equal to ULN for the lab.
* Urine protein/creatinine (UPC) ratio must be less than 1.0.
* All patients must have their LVEF assessed by 2-D echocardiogram within 3 months prior to study entry. (MUGA scan may be substituted for 2-D echocardiogram based on institutional preferences.) The LVEF must be greater than/equal to 55% regardless of the institution's LLN.
* Note: Since the pre-entry LVEF serves as the baseline for comparing subsequent LVEF assessments to determine if trastuzumab and bevacizumab therapy can be administered, it is critical that this baseline study be an accurate assessment of the patient's LVEF. If the baseline LVEF is greater than 65%, the investigator is encouraged to have the accuracy of the initial LVEF result confirmed and to consider repeating the study if the accuracy is uncertain.

Exclusion Criteria:

Conditions for patient ineligibility (Cohort A)

* FNA alone to diagnose the primary tumor.
* Surgical axillary staging procedure prior to study entry. (Procedures that are permitted include: 1) FNA or core biopsy of an axillary node for any patient, and 2) although not recommended, a pre-neoadjuvant therapy SN biopsy for patients with clinically negative axillary nodes.

Condition for patient ineligibility (Cohort B)

• Breast reconstruction using tissue expanders or implants at the time of mastectomy.

Conditions for patient ineligibility (ALL patients)

* Definitive clinical or radiologic evidence of metastatic disease.
* Synchronous bilateral invasive breast cancer.
* History of ipsilateral or contralateral invasive breast cancer regardless of treatment or ipsilateral DCIS treated with RT.
* History of non-breast malignancies within the 5 years prior to study entry. Patients with the following cancers are eligible if diagnosed and treated within the previous 5 years: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.
* Prior therapy with anthracyclines, taxanes, trastuzumab, or bevacizumab for any malignancy.
* Treatment including RT, chemotherapy, and/or targeted therapy, administered for the currently diagnosed breast cancer prior to study entry.
* Continued therapy with any hormonal agent such as raloxifene, tamoxifen, or other SERM. (Patients are eligible if these medications are discontinued prior to study entry.)
* Any sex hormonal therapy, e.g., birth control pills, ovarian hormone replacement therapy, etc. These patients are eligible if this therapy is discontinued prior to study entry. (Women of reproductive potential must agree to use an effective non-hormonal method of contraception during study therapy and for at least 6 months after completion of targeted therapy.)
* Cardiac disease that would preclude the use of the drugs included in the FB-5 treatment regimen. This includes but is not confined to:

  * Active cardiac disease: angina pectoris that requires the use of anti-anginal medication; ventricular arrhythmias except for benign premature ventricular contractions controlled by medication; supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication; conduction abnormality requiring a pacemaker; and clinically significant valvular disease.
  * History of cardiac disease: myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LV function; documented CHF; or documented cardiomyopathy.
* Uncontrolled hypertension defined as systolic BP greater than 150 mmHg or diastolic BP greater han 90 mmHg, with or without anti-hypertensive medication. Patients with initial BP elevations are eligible if initiation or adjustment of BP medication lowers pressure to meet entry criteria.
* History of hypertensive crisis or hypertensive encephalopathy.
* History of TIA or CVA.
* History of other arterial thrombotic event within 12 months before study entry.
* Symptomatic peripheral vascular disease.
* Any significant bleeding within 6 months before study entry, exclusive of menorrhagia in premenopausal women.
* Serious or non-healing wound, skin ulcers, or bone fracture.
* Gastroduodenal ulcer(s) determined by endoscopy to be active.
* History of GI perforation, abdominal fistulae, or intra-abdominal abscess.
* Anticipation of need for major surgical procedures (other than the breast surgery required for patients in Cohort A) during study therapy and for at least 3 months following completion of bevacizumab.
* Known bleeding diathesis, coagulopathy, or requirement for therapeutic doses of coumadin.
* Other nonmalignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow-up.
* Sensory/motor neuropathy greater than/equal to grade 2, as defined by the NCI's CTCAE v3.0.
* Conditions that would prohibit administration of corticosteroids.
* History of hypersensitivity reaction to drugs formulated with polysorbate 80.
* Pregnancy or lactation at the time of study entry. (Note: Pregnancy testing should be performed according to institutional standards for women of child-bearing potential.)
* Use of any investigational agent within 4 weeks prior to enrollment in the study.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2007-05; Primary Completion 2009-12 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (36):
- United States (35):
  - Clearview Cancer Institute- Huntsville, Huntsville, Alabama
  - Kaiser Permanente-San Diego, San Diego, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - CCOP, Colorado Cancer Research Program, Inc., Denver, Colorado
  - Baptist Regional Cancer Institute, Jacksonville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - CCOP, Central Illinois, Springfield, Illinois
  - CCOP, Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - University of Iowa, Iowa City, Iowa
  - NortonHealtcare Inc., Louisville, Kentucky
  - CCOP, Grand Rapids Clnical Oncology Program, Grand Rapids, Michigan
  - CCOP, Michigan Cancer Research Consortium, Grosse Pointe Woods, Michigan
  - CCOP, Kalamazoo, MI, Kalamazoo, Michigan
  - Michigan State University - Breslin Cancer Center, Lansing, Michigan
  - CCOP, Metro-Minnesota, Minneapolis, Minnesota
  - CCOP, Cancer Research for the Ozarks, Springfield, Missouri
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University Hospital and Medical Center - SUNY, Stony Brook, New York
  - CCOP, Southeast Cancer Control Consortium, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Case Western Reserve/University Hospitals-Ireland Cancer Cntr., Cleveland, Ohio
  - CCOP, Dayton, OH, Dayton, Ohio
  - CCOP, Columbia River Oncology, Portland, Oregon
  - Kimmel Cancer Center at Jefferson, Philadelphia, Pennsylvania
  - Albert Einstein Healthcare Network, Philadelphia, Pennsylvania
  - Allegheny General Hospital/Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - NSABP Foundation, Inc., Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - CCOP, Upstate Carolina, Spartanburg, South Carolina
  - Joe Arrington Cancer Research & Treatment Center, Lubbock, Texas
  - CCOP, Scott and White Memorial Hospital, Temple, Texas
  - MBCCOP, Virginia Commonwealth University, Richmond, Virginia
  - CCOP, Marshfield Clinic, Marshfield, Wisconsin
- University of Montreal Hospital Group, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: • Cohort A: Women with unresected locally advanced breast cancer (clinical Stage IIIA, IIIB, and IIIC)
- Cohort B: • Cohort B: Women with resected pN2 or pN3 (pathologic Stage III) breast cancer
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 76 | 29
Completed | 76 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 76 | 29 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (9.6) | 53.8 (11.4) | 49.7 (10.4)
Age, Customized [Number; unit: participants]
  18 to less than 50 years | 39 | 10 | 49
  >=50 years and <=59 years | 27 | 8 | 35
  > 59 years | 10 | 11 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 29 | 105
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 65 | 26 | 91
  Black or African American | 10 | 3 | 13
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  American Indian or Alaskan Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Unknown | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 70 | 29 | 99
  Unknown | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Pathological Complete Response (pCR) in the Breast and Nodes for Patients With HER2-positive LABC Following Neoadjuvant Treatment (Cohort A)
Description: The determination of pCR is performed by the local pathologist following examination of tissue (breast and nodes)removed at the time of surgery. The outcome measure is the number of participants with no histologic evidence of invasive tumor cells in the surgical breast specimen, axillary nodes, or SNs identified after neoadjuvant chemotherapy.
Time Frame: Assessed at time of surgery on average at 8 months
Population: 73 of the 76 patients in Cohort A were analyzed: 2 patients did not have surgery and 1 patient did not have the nodal status determined.
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 73 | 0
participants | 34 [34.8 to 58.63] |

2. Primary Outcome: Number of Participants With Cardiac Events
Description: The number of cardiac events defined as NYHA Class III/IV CHF and cardiac death.To determine the rate of cardiac events (NYHA Class III/IV CHF and cardiac death) of a regimen of EC followed by THA when administered to: Cohort A as neoadjuvant therapy for HER-2 positive locally advanced (clinical stage IIIA, IIIB or IIIC breast cancer or Cohort B as adjuvant therapy for resected HER2-positive pN2 or pN3 (pathologic stage III) breast cancer. The number of participants with one or more cardiac events are being reported.
Time Frame: Cohort A: Baseline, post-treatment with EC, 2-4 weeks after surgery, and 9, 12, 15, and 18 months from study entry. Cohort B: Baseline, post-treatment with EC, 2-3 weeks after the last dose of docetaxel, and 6, 9, 12, 15, and 18 months from study entry.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 70 | 29
Participants | 4 | 0

3. Secondary Outcome: Number of Participants With no Histologic Evidence of Invasive Tumor Cells in the Surgical Breast Specimen.
Description: The determination of pCR will be performed by the local pathologist following examination of tissue (breast and nodes) removed at the time of surgery.
Time Frame: Assessed at the time of surgery
Population: Endpoint was for Cohort A only.70
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 70 | 0
Participants | 36 | 0

4. Secondary Outcome: Clinical Complete Response (cCR)
Description: cCR following the last dose of docetaxel (Cohort A). cCR is detemined by tumor measurement by physical exam at baseline: target lesions greater than or equal to 2.0 cm; non-target lesions greater than or equal to 2.0 cm. cCR assessment at other timepoints: resolution of all target and non-target lesions identified at baseline, and no new lesions or other signs of disease progression.
Time Frame: Determined at baseline, 2-3 weeks after the last EC dose, 2-4 weeks after last Docetaxel dose-before surgery.
Population: This outcome only applicable to Cohort A.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Cohort A: * Cohort A: Women with unresected locally advanced breast cancer (clinical Stage IIIA, IIIB, and IIIC)
  * Cohort B: Women with resected pN2 or pN3 (pathologic Stage III) breast cancer
  Epirubicin: Both Cohorts: Epirubicin 90 mg/m2 IV every 21 days x 4 cycles
  Cyclophosphamide: Both Cohorts: Cyclophosphamide 600 mg/m2 IV every 21 days x 4 cycles
  Docetaxel: Both Cohorts: Docetaxel 100 mg/m2 IV on Day 1 every 21 days x 4 cycles
  Trastuzumab: Cohort A: Pre-op therapy - 4 mg/kg IV first dose, then subsequent doses at 2 mg/kg IV weekly (16+ weeks) until 1-7 days prior to surgery. Post-operative therapy (beginning no sooner than 28 days after surgery and continuing every 3 weeks x 13 doses) - 8 mg/kg IV first post-op dose, then subsequent doses at 6 mg/kg IV
  Cohort B: 4 mg/kg IV first dose, then subsequent doses at 2 mg/kg IV weekly on days 1, 8, and 15. Three (3) weeks after last dose of docetaxel, 6 mg/kg IV and continuing every 3 weeks x 13 doses
  Bevacizumab: Cohort A: Cycles 1-4, 15 mg/kg IV on day 1 of cycle 4 only; Cycles 5-7, 15 mg/kg IV on day 1 every 21 days x 3 cycles; post-operative therapy (beginning no sooner than 28 days after surgery), 15 mg/kg IV every 3 weeks x 13 doses
  Cohort B: Cycles 5-8, 15 mg/kg IV on day 1 every 21 days x 4 cycles; beginning 3 weeks after last dose of docetaxel, 15 mg/kg IV every 3 weeks x 13 doses
Arm/Group | Cohort A
Number analyzed (Participants) | 70
percentage of patients | 61.43 [49.03 to 72.83]

5. Secondary Outcome: Grade 3 and 4 Toxicities, Including Toxicities Associated With Radiation Therapy(RT)
Time Frame: Before each cycle of pre-op Rx; 2-4 wks after the last docetaxel dose; 2-4 wks post surgery (Cohort A); every 6 wks during post-op Rx (Cohort A); every 6 wks during targeted therapy alone (Cohort B); RT complications assessed at 12 mos from study entry
Population: Data shows total number of patients with 1 AE, for further information see Reported Adverse Events Section.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 76 | 29
Participants | 55 | 22

6. Secondary Outcome: Recurrence-free Survival
Description: To determine the five-year RFS.
Time Frame: From the first dose of study therapy until the date of recurrence or for a maximum of five (5) years from study entry
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 70 | 29
percentage of patients | 75.97 [63.5 to 85.67] | 89.66 [71.2 to 96.54]

7. Secondary Outcome: Overall Survival
Description: Death from any cause during the 5 years from study entry.
Time Frame: From the first dose of study therapy until the date of death or for a maximum of five (5) years from study entry
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 76 | 29
Participants | 12 | 0

8. Secondary Outcome: Percentage of Participants With Surgical Complications (From Mastectomy, Lumpectomy, and Axillary Staging Procedures) (Cohort A)
Description: The percentage of patients with surgical complications (from mastectomy, lumpectomy, and axillary staging procedures).
Time Frame: 2-4 weeks after surgery and at 9 and 12 months from study entry
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A
Number analyzed (Participants) | 74
Participants | 37

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Cohort A | Cohort B
Serious Adverse Events (participants affected / at risk) | 16/76 | 5/29
Other Adverse Events (participants affected / at risk) | 76/76 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=76) | Cohort B (N=29)
Pain- head/headache (General disorders) | 3 | 0
Pain- back (General disorders) | 2 | 0
Pain- extremity-limb (General disorders) | 1 | 0
Pain- joint (General disorders) | 1 | 0
Pain- NOS (General disorders) | 1 | 0
Pain- chest/thorax (General disorders) | 0 | 1
Infection with normal ANC - skin (cellulites) (Infections and infestations) | 2 | 1
Infection with Normal ANC - bladder (urinary) (Infections and infestations) | 1 | 0
Dehydration (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Creatinine (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Left ventricular systolic function (Cardiac disorders) | 1 | 0
Hypertension (Cardiac disorders) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1
Hemorrhage, GI - stomach (Gastrointestinal disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 1 | 0
Syncope (General disorders) | 2 | 1
Mood alteration - depression (Psychiatric disorders) | 2 | 0
Pain - neck (General disorders) | 2 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypertriglyceridemia (Investigations) | 1 | 0
Infection documented clinically or micro with grade 4 neutrophils - blood (Infections and infestations) | 1 | 0
Infection with unknown ANC - wound (Infections and infestations) | 1 | 0
Infection other - colon (Infections and infestations) | 1 | 0
Infection other - skin (cellulitis) (Infections and infestations) | 1 | 0
Myositis (General disorders) | 1 | 0
Neurology - other - loss of consciousness (Nervous system disorders) | 1 | 0
Perforation, GI - colon (Gastrointestinal disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Hemorrhage pulmonary - nose (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ulcer, GI - stomach (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=76) | Cohort B (N=29)
Alopecia (Skin and subcutaneous tissue disorders) | 65 | 24
Rash (Skin and subcutaneous tissue disorders) | 13 | 9
Hand - foot (Skin and subcutaneous tissue disorders) | 9 | 2
Pain - muscle (General disorders) | 28 | 11
Pain - bone (General disorders) | 25 | 14
Pain - joint (General disorders) | 19 | 12
Pain - head/headache (General disorders) | 19 | 6
Pain - extremity - limb (General disorders) | 16 | 4
Pain - chest/thorax (General disorders) | 11 | 2
Pain - breast (General disorders) | 9 | 1
Pain - back (General disorders) | 8 | 6
Pain - abdominal NOS (General disorders) | 8 | 2
Pain - pain NOS (General disorders) | 5 | 6
Mucositis (functional/symptomatic) - oral cavity (Gastrointestinal disorders) | 31 | 8
Vomiting (Gastrointestinal disorders) | 24 | 7
Nausea (General disorders) | 23 | 12
Diarrhea (Gastrointestinal disorders) | 17 | 6
Dehydration (Gastrointestinal disorders) | 15 | 7
Constipation (Gastrointestinal disorders) | 10 | 1
Heartburn (Gastrointestinal disorders) | 9 | 2
Fatigue (General disorders) | 47 | 20
Fever (General disorders) | 4 | 1
Hypertension (Cardiac disorders) | 29 | 12
Left ventricular systolic function (Cardiac disorders) | 13 | 3
Neutrophils (Blood and lymphatic system disorders) | 19 | 5
Leucocytes (Blood and lymphatic system disorders) | 17 | 3
Hemoglobin (Blood and lymphatic system disorders) | 10 | 7
Neuropathy - sensory (Nervous system disorders) | 18 | 8
Dizziness (Nervous system disorders) | 6 | 1
Neuropathy - motor (Nervous system disorders) | 5 | 1
Infection with normal ANC - skin (cellulites) (Infections and infestations) | 11 | 1
Infection with normal ANC - bladder (urinary) (Infections and infestations) | 6 | 6
Febrile neutropenia (Infections and infestations) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 1
ALT (Metabolism and nutrition disorders) | 4 | 1
AST, SGOT (Metabolism and nutrition disorders) | 4 | 1
Nail Changes (Skin and subcutaneous tissue disorders) | 16 | 9
Hot flashes (General disorders) | 15 | 4
Mucositis (clinical exam) - oral cavity (Gastrointestinal disorders) | 14 | 5
Lymphopenia (Blood and lymphatic system disorders) | 12 | 7
Anorexia (General disorders) | 12 | 5
Taste alteration (Gastrointestinal disorders) | 12 | 4
Mood alteration - depression (Psychiatric disorders) | 11 | 5
Insomnia (General disorders) | 10 | 3
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Mood alteration - anxiety (Psychiatric disorders) | 9 | 1
Edema - limb (General disorders) | 6 | 1
Gastritis (Gastrointestinal disorders) | 6 | 0
Watery eye (Eye disorders) | 5 | 6
Weight loss (General disorders) | 5 | 3
Hyperglycemia (Investigations) | 5 | 1
Tinnitus (Ear and labyrinth disorders) | 5 | 1
Infection with normal ANC - sinus (Infections and infestations) | 5 | 0
Infection with unknown ANC - sinus (Infections and infestations) | 5 | 0
Infection with unknown ANC - upper airway NOS (Infections and infestations) | 5 | 0
Esophagitis (Gastrointestinal disorders) | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Infection with normal ANC - upper airway NOS (Infections and infestations) | 3 | 2
Infection with unknown ANC - bronchus (Infections and infestations) | 3 | 2
Blurred vision (Eye disorders) | 2 | 3
Hemorhoids (Gastrointestinal disorders) | 1 | 5
Hyponatremia (Metabolism and nutrition disorders) | 2 | 2
Blood - Other (low HCT) (Blood and lymphatic system disorders) | 4 | 0
Vaginitis (Reproductive system and breast disorders) | 2 | 2
Infection - other- shingles (Infections and infestations) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less